CLINICAL TRIAL: NCT00882895
Title: Autologous Followed by Non-myeloablative Allogeneic Transplantation for Non-Hodgkin's Lymphoma
Brief Title: Tandem Stem Cell Transplantation for Non-Hodgkin's Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0042 / 201101864
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Lymphoma, Non-Hodgkin; Transplantation, Autologous; Transplantation, Homologous; Total Lymphoid Irradiation; Anti-thymocyte globulin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Antilymphocyte Serum; thymoglobulin; Methylprednisolone Hemisuccinate; Methylprednisolone; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Allogeneic Transplant (Experimental): * TLI - 80 cGy on days -14, -11, -10, -9, -8, -7, -4, -3, -2, -1
  * Anti-thymocyte globulin (ATG) 1.5 mg/kg on days -11, -10, -8, -7
  * Solumedrol - 1 mg/kg on days -11, -10, -9, -8, -7
  * Tacrolimus - beginning on day -3 with starting dose of 0.3 mg/kg PO BID. Will be continued per institutional guidelines.
  * Stem cell infusion - day 0
  * Mycophenolate mofetil (MMF) - beginning on day 0 with dose of 15 mg/kg PO (5-10 hours after transplant)
  Interventions: Procedure: Stem cell infusion; Procedure: TLI; Drug: Anti-thymocyte globulin; Drug: Solumedrol; Drug: Tacrolimus; Drug: Mycophenolate mofetil

INTERVENTIONS:
Procedure: Stem cell infusion
Procedure: TLI
Drug: Anti-thymocyte globulin
  Other Names: ATG; Atgam; Thymoglobulin
Drug: Solumedrol
  Other Names: Medrol; Solu-Medrol
Drug: Tacrolimus
  Other Names: FK-506; Prograf; Advagraf; Protopic
Drug: Mycophenolate mofetil
  Other Names: MMF; CellCept; Myfortic

SUMMARY:
This is a research study testing a new approach to treating high-risk non-Hodgkin's lymphoma consisting of an autologous hematopoietic (blood) stem cell transplant (using a patient's own hematopoietic cells) followed by a non-myeloablative allogeneic transplantation (transplant from another individual).

The investigators hypothesize that the addition of the second non-myeloablative transplant will improve the chances for long-term control of lymphoma.

DETAILED DESCRIPTION:
The approach to recurrent or primary refractory non-Hodgkin's lymphoma has been to treat patients with second-line chemotherapy (usually 2-3 courses) for the purposes of cytoreduction and to establish sensitivity to chemotherapy. Thereafter, peripheral blood progenitor cells have been mobilized with cyclophosphamide and granulocyte colony stimulating factor, apheresed and cryopreserved. Unfortunately, there are subgroups of patients with poor outcomes using autologous transplantation including those with transformed lymphoma as well as patients who do not attain a minimal disease state due to chemoresistant disease.

In a group of 17 patients with transformed lymphoma who received autologous transplants at Stanford University, the median EFS and OS were 1.48 and 2.7 years respectively with a 7-year survival of only 20%. In comparison, patients with chemosensitive follicular lymphoma who received the same regimen also had a poor median EFS of 1.3 years, but the median survival was 6.7 years. The outcomes for patients with chemotherapy-resistant relapsed NHL is also poor with EFS in the range of 20% in many studies of autologous transplantation.

These groups of patients have limited disease control and survival with standard chemotherapy regimens, and although they often have excellent cytoreduction with the high-dose chemotherapy regimen, relapse remains the primary cause of treatment failure. The current trial utilizes a similar approach that we have taken with patients with multiple myeloma, who appear to benefit from an allogeneic graft-versus-tumor effect, using a combined autologous and non-myeloablative allogeneic transplant regimen to reduce transplant-related complications. In addition, there are limited reports of using an autologous/allogeneic approach for lymphoma patients using non-myeloablative allogeneic transplants. Eligible patients will be treated with high-dose chemotherapy using BCNU, etoposide, cytarabine and melphalan with autologous hematopoietic cell support as a method of cytoreduction. Approximately 60-120 days after the autologous transplant, patients will receive an allogeneic transplant using a preparative regimen of total lymphoid irradiation and anti-thymocyte globulin in an attempt to develop a graft-versus-lymphoma effect.

ELIGIBILITY:
Inclusion Criteria

* Age 18 to 70 years.
* Histologically proven non-Hodgkin's lymphoma
* High risk disease including at least one of the following:

  * Relapsed or refractory disease
  * Transformed lymphoma
  * Aggressive T-cell lymphoma
  * Failure to achieve completed remission (CR) following Auto SCT
  * Less than a 20% chance of event-free survival from autologous transplant determined by the treating physician and the Principal Investigator
* ECOG performance status < or = 2
* Underwent Autologous SCT 60-120 days prior to registration including:

  * BEAM conditioning (BCNU: 300 mg/m2 IV day -7, Etoposide: 100 mg/m2 IV BID days -6,-5,-4,-3, Cytarabine: 100 mg/m2 IV BID days -6,-5,-4,-3, Melphalan: 140 mg/m2 IV day -2)
  * Minimum of 2 x 106 CD34+ cells/kg infused
* Full hematologic recovery following Auto HCT including:

  * Absolute neutrophil count (ANC) >1000 µl
  * Platelet count of ≥50,000 µl independent of transfusion for >7 days
* Available matched related or unrelated donor. Selected donor must be a complete match or have only a single antigen mismatch.
* Women of child-bearing potential and sexually active males must use an accepted and effective method of birth control.
* Bone marrow comprising of < 10% lymphoma on most recent biopsy/aspiration (within 9 months of Allo transplant; may have been performed prior to autologous transplant).
* Serum bilirubin < or = 2 x the institutional ULN
* Serum creatinine < or = 2 x the institutional ULN and measured or estimated creatinine clearance > 60 cc/min by the following formula

  * Estimated Creatinine Clearance = (140 age)X WT(kg) X 0.85 if female 72X serum creatinine(mg/dl).
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria

* Prior autologous or allogeneic hematopoietic cell transplantation (other than autologous SCT 60-120 days prior to registration)
* Prior radioimmunotherapy
* Known or suspected progressive disease following autologous SCT
* Additional treatment for NHL administered from time of autologous SCT through registration
* Pregnant or breast-feeding women (due to the known birth defects association with the treatments used in this study)
* Human immunodeficiency virus (HIV)-positive (the concern for opportunistic infection and hematologic reserve are considered to be significantly greater in this population.)
* Any prior malignancy is allowed except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or other cancer for which the patients has been disease-free for five years.
* Active infection requiring oral or intravenous antibiotics.

Inclusion of Women and Minorities

-Both men and women and members of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-05-05 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Determine the event free survival | Up to 10 years from transplant
Determine the toxicities | Day 100

SECONDARY OUTCOMES:
To evaluate the kinetics of donor hematopoietic cell engraftment and chimerism. | Day 56, Day 100, Day 180, and Day 365
To evaluate the incidence and extent of acute and chronic GVHD. | Up to 10 years
To evaluate the overall and non-relapse mortality rate. | Up to 10 years
Incidence of chemotherapy-associated pneumonitis | Day 100

CONTACTS AND LOCATIONS:
Overall Officials: Keith Stockerl-Goldstein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maloney DG, Molina AJ, Sahebi F, Stockerl-Goldstein KE, Sandmaier BM, Bensinger W, Storer B, Hegenbart U, Somlo G, Chauncey T, Bruno B, Appelbaum FR, Blume KG, Forman SJ, McSweeney P, Storb R. Allografting with nonmyeloablative conditioning following cytoreductive autografts for the treatment of patients with multiple myeloma. Blood. 2003 Nov 1;102(9):3447-54. doi: 10.1182/blood-2002-09-2955. Epub 2003 Jul 10. PMID 12855572
- See also: Alvin J. Siteman Cancer Center at Barnes Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu